CLINICAL TRIAL: NCT04283110
Title: Impact of Adding Midzolam to Bupavicaine 0.5% in Regional Spinal Anaesthesia on Maternal Middle Cerebral Artery Velocimetry in Parturients With Severer Preeclampsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mina Maher, dr, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 293:9/2019
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Midazolam in Preeclamptic Patients

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam group (Active Comparator): Midazolam group will receive 1 mg intrathecal midazolam once during induction for anethesia
  Interventions: Drug: intrthecl midazolam
- control group (No Intervention): control group will receive placebo ( 0.5cm of sterile saline

INTERVENTIONS:
Drug: intrthecl midazolam — midazolm as as adjuvant in spinal anesthesia
  Arms: Midazolam group

SUMMARY:
Trial to use GABA mimetic action of midazolam to ameliorate the severe preeclampsia induced neuronal excitotoxicity using middle cerebral artery transcranial doppler resisitive vasculer indices to evaluate . Secondery goal is to study end organ injury

ELIGIBILITY:
Inclusion Criteria:

* All parturients with severe preeclampsia for urgent C.S

Exclusion Criteria:

* Ladies refusal to participate. Refusal to have spinal anesthsia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — All cases are ladies with severe preeclampsia
Enrollment: 100 (Estimated)
Dates: Start 2019-01-12 (Actual); Primary Completion 2020-02-17 (Estimated); Study Completion 2020-04-05 (Estimated)

PRIMARY OUTCOMES:
Measuring Pulsatality index and resistive index of maternal middle cerebral artery | 2 months
  Resistive vasculer indices outcome after intrthecal midazolam injection

CONTACTS AND LOCATIONS:
Locations (1):
- Elminia university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
All data of primary and secondery outcome measures will be avaliable